CLINICAL TRIAL: NCT03690557
Title: Examining Reach and Implementation of an Evidence-based Weight Loss Program in Rural Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0581-18-EP
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: Delivery of Health Care; Rural Health; Primary Health Care; Outcomes and Process Assessment (Health Care)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IncentaHealth (Experimental): All patients who decide to join the weight loss program will be enrolled in the commercially-available IncentaHealth program - a comprehensive, evidence-based, behavioral weight management program designed to help patients initiate and maintain weight loss. The program is delivered completely online, via website, emails, mobile app, and (if requested by the participant) text messaging over 12 months. Each participant will be given a digital scale that wirelessly syncs with a smartphone app. Participants' weights are automatically uploaded to the Incentahealth online portal. In the informed consent process, participants will need to agree to release their weight data to researchers at the University of Nebraska Medical Center in order to participate in this program.
  Interventions: Behavioral: IncentaHealth

INTERVENTIONS:
Behavioral: IncentaHealth — IncentaHealth is a comprehensive, behavioral weight management program designed to help individuals initiate and maintain weight loss. Individuals participate in the IncentaHealth program from their homes, receive program information electronically through daily emails and through a smartphone app for the duration of the study, and have the option to receive text messages and speak with health coaches over the telephone. Participants in this study will be enrolled in the IncentaHealth program for 12 months, and will engage with health coaching, tracking of body weight, and are provided a number of resources for healthy living throughout the 12 months.

SUMMARY:
The majority of American adults do not meet recommended guidelines for healthy eating or physical activity and are overweight or obese, which puts them at risk for chronic disease, poor quality of life, and increased personal and public health care costs. Despite the development and success of a number of evidence-based weight management interventions, these programs have lacked systematic and consistent translation in clinical practice or community services. Further, few of these interventions have been tested in rural populations, where there is a disproportionally high number of obese individuals, and resources to support such programs are lacking. Primary care clinics have the necessary resources to support such programs, and might be the ideal setting to intervene and address concerns of weight loss and management in rural areas. The intent of the proposed project is to increase the capacity of primary care in rural Nebraska to translate evidence-based weight management approaches into practice, improve the speed of uptake and the likelihood of sustainability, and reach a large and representative group of individuals. To achieve this, the investigators will 1) conduct a limited effectiveness and feasibility study to determine impact on weight loss of 100 overweight and obese adult patients in a rural Nebraska primary care clinic, and 2) test multiple strategies for recruitment to determine best practices for program reach. The primary outcome for program effectiveness is percent body weight loss, and the primary outcome for program feasibility is reach, defined as the proportion of individuals who enroll in the program per each recruitment strategy. The proposed project provides a means of implementing an evidence-based weight loss program in rural Nebraska, has the capacity to create meaningful change in patient weight status, and has the potential to influence future efforts to translate evidence-based weight management programs into rural primary care practice.

DETAILED DESCRIPTION:
In the United States, the choice to eat energy-dense foods and engage in sedentary activities is attractive and convenient. More than two thirds of adults in the US are either overweight or obese, with rural residents experiencing a disproportionally higher prevalence of obesity, particularly in the state of Nebraska. Excess body weight carries with it a host of adverse conditions: type II diabetes, coronary heart disease, hypertension, some cancers, and early mortality. The high prevalence of obesity and its consequences have catalyzed the development of many weight management interventions that have been effective in helping individuals initiate weight loss and maintain a healthy weight. Despite their demonstrated efficacy, few of these programs have been systematically and consistently translated into typical clinical practice or community services. This translation is especially scarce in rural communities.

Programs designed to improve weight loss that target rural communities can be a challenge to design and implement, due to the lack of resources available in rural communities to support such programs. However, primary care clinics may provide an ideal setting to implement effective diet, physical activity, and weight management support. Despite the lack of resources, most rural communities have a primary care provider who is trusted by patients to provide counseling on healthy behaviors. Furthermore, programs delivered through the private sector that engage patients and organizational decision makers, such as primary care providers, are hypothesized to be more sustainable.

Primary care systems may offer a practical and sustainable method of implementing meaningful weight management interventions, but few weight management programs are currently available that can be readily adopted into rural primary care practice. To address the gap in translating programs into practice, the investigators will use the National Cancer Institutes (NCI) Putting Public Health Evidence in Action process, which provides steps for defining evidence-based programs, assessing resources and need in the community, and ultimately choosing an evidence based program for implementation. The investigators will modify the NCI process to include, but move beyond, simply considering the magnitude of weight loss as the primary factor in the selection process. Additionally, the investigators will address factors related to scalability, clinical uptake, and sustainability which are key for the translation of evidence-based interventions into practice. The RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) framework will be used to consider the impact at the individual and organizational levels of the weight management approaches. Reach (i.e., the participation rate of individuals from the target population and representativeness of those who participate) and effectiveness are the two factors considered to contribute to overall impact when translating evidence-based strategies into typical practice. These factors can be addressed by developing a system within primary care that provides opportunities for quick and representative accrual of participants, provides clinics with an evidence-based program, and provides a tracking and evaluating system to determine the potential population health impact of the intervention.

The intent of the proposed project is to increase the capacity of primary care in rural Nebraska to translate evidence-based weight management approaches into practice, improve the speed of uptake and the likelihood of sustainability, and reach a large and representative group of individuals.Effective weight loss programs are available, but the question of how best to deliver these interventions to the general public remains. The proposed study will help to improve the translation of evidence-based programs into typical clinical practice and determine best practices for patient recruitment and referral. This will be done through the completion of the following aims:

Aim 1: Conduct a limited effectiveness and feasibility (including cost) study of the IncentaHealth intervention to determine impact on weight loss of 100 overweight and obese patients. The proportion of participants who experience a clinically meaningful weight loss (i.e., 5% initial body weight) at 6-months and cost per participant achieving this bench march will also be reported.

Aim 2: Test methods to increase intervention reach using a 2X2 randomized recruitment design (in-visit referral vs electronic health record screening and mailed referral; active vs passive follow-up) within a rural primary care clinic in Nebraska.

The completion of these aims has the potential to affect the health of rural Nebraskans and influence future efforts to translate evidence-based weight management programs into rural primary-care practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of Butler County Clinic in David City, Nebraska
2. BMI ≥25 (determined by patients electronic medical record measurement)
3. Aged 19 or older
4. Own an Apple or Android smartphone
5. Have an active email address and have an understanding of how to navigate the internet
6. Able to engage in physical activity and modify eating habits
7. Approved to participate by primary care provider
8. Capable of providing consent to participate

Exclusion Criteria:

1. Not meeting all inclusion criteria
2. Currently scheduled for bariatric surgery or had bariatric surgery within the past 3 years
3. Currently undergoing treatment for cancer
4. Currently on a prescribed medical diet
5. Diagnosed with an eating disorder
6. Currently participating in another weight management activity or interventional research trial
7. Had a heart attack or stroke within the past 6 months or currently in cardiac rehabilitation
8. Currently on dialysis or an active organ transplant list
9. Currently pregnant or planning to become pregnant in the next 12 months
10. Planning to move outside of the recruitment area in the next 12 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Percent of Initial Body Weight Lost/Gained [Effectiveness] | Baseline, 6, and 12 months
  Change in weight, measured in percent of body weight
Enrollment Rate per Each Recruitment Strategy [Reach] | In two-week intervals until recruitment cap is met
  Proportion of individuals who enroll in the program per each recruitment strategy

SECONDARY OUTCOMES:
Clinically Meaningful Weight Loss | Baseline, 6, and 12 months
  Yes/no did the participant lose 5% of their initial body weight

OTHER OUTCOMES:
Change in Weight Loss Self-Efficacy Questionnaire Scores | Baseline and 12 months
  Changes in scores of self-efficacy for weight loss using the Weight Loss Self-Efficacy subscale as described in Wilson et al, 2016. Scores range from 0 (least confident) to 100 (most confident). An increase in score from baseline to 12 months indicates an increase in self-efficacy for weight loss.
Change in Physical Activity Self-Efficacy Questionnaire Scores | Baseline and 12 months
  Changes in scores of self-efficacy for physical activity using the Physical Activity Self-Efficacy subscale as described in Wilson et al, 2016. Scores range from 0 (least confident) to 100 (most confident). An increase in score from baseline to 12 months indicates an increase in self-efficacy for physical activity.
Change in Healthful Eating Self-Efficacy Questionnaire Scores | Baseline and 12 months
  Changes in scores of self-efficacy for healthful eating using the Healthful Eating Self-Efficacy subscale as described in Wilson et al, 2016. Scores range from 0 (least confident) to 100 (most confident). An increase in score from baseline to 12 months indicates an increase in self-efficacy for healthful eating.

CONTACTS AND LOCATIONS:
Overall Officials: Gwenndolyn C Porter, MS, Principal Investigator — University of Nebraska
Locations (1):
- Butler County Clinic, David City, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Befort CA, Nazir N, Perri MG. Prevalence of obesity among adults from rural and urban areas of the United States: findings from NHANES (2005-2008). J Rural Health. 2012 Fall;28(4):392-7. doi: 10.1111/j.1748-0361.2012.00411.x. Epub 2012 May 31. PMID 23083085
- [Background] Perri MG, Limacher MC, Durning PE, Janicke DM, Lutes LD, Bobroff LB, Dale MS, Daniels MJ, Radcliff TA, Martin AD. Extended-care programs for weight management in rural communities: the treatment of obesity in underserved rural settings (TOURS) randomized trial. Arch Intern Med. 2008 Nov 24;168(21):2347-54. doi: 10.1001/archinte.168.21.2347. PMID 19029500
- [Background] Perri MG, Sears SF Jr, Clark JE. Strategies for improving maintenance of weight loss. Toward a continuous care model of obesity management. Diabetes Care. 1993 Jan;16(1):200-9. doi: 10.2337/diacare.16.1.200. PMID 8422776
- [Background] Perri MG, McAdoo WG, Spevak PA, Newlin DB. Effect of a multicomponent maintenance program on long-term weight loss. J Consult Clin Psychol. 1984 Jun;52(3):480-1. doi: 10.1037//0022-006x.52.3.480. No abstract available. PMID 6747068
- [Background] Glasgow RE, Goldstein MG, Ockene JK, Pronk NP. Translating what we have learned into practice. Principles and hypotheses for interventions addressing multiple behaviors in primary care. Am J Prev Med. 2004 Aug;27(2 Suppl):88-101. doi: 10.1016/j.amepre.2004.04.019. PMID 15275677
- [Background] Ely AC, Befort C, Banitt A, Gibson C, Sullivan D. A qualitative assessment of weight control among rural Kansas women. J Nutr Educ Behav. 2009 May-Jun;41(3):207-11. doi: 10.1016/j.jneb.2008.04.355. PMID 19411055
- [Background] Ard JD. Unique perspectives on the obesogenic environment. J Gen Intern Med. 2007 Jul;22(7):1058-60. doi: 10.1007/s11606-007-0243-z. No abstract available. PMID 17520309
- [Background] Swinburn B, Egger G. The runaway weight gain train: too many accelerators, not enough brakes. BMJ. 2004 Sep 25;329(7468):736-9. doi: 10.1136/bmj.329.7468.736. PMID 15388619
- [Background] Rural 2010 Health Goals and Objectives for Nebraska: Progress Report.; 2008. http://dhhs.ne.gov/Documents/Rural_Prog_Rpt.pdf. Accessed July 21, 2016.
- [Background] Guh DP, Zhang W, Bansback N, Amarsi Z, Birmingham CL, Anis AH. The incidence of co-morbidities related to obesity and overweight: a systematic review and meta-analysis. BMC Public Health. 2009 Mar 25;9:88. doi: 10.1186/1471-2458-9-88. PMID 19320986
- [Background] Olshansky SJ, Passaro DJ, Hershow RC, Layden J, Carnes BA, Brody J, Hayflick L, Butler RN, Allison DB, Ludwig DS. A potential decline in life expectancy in the United States in the 21st century. N Engl J Med. 2005 Mar 17;352(11):1138-45. doi: 10.1056/NEJMsr043743. PMID 15784668
- [Background] Donnelly JE, Hill JO, Jacobsen DJ, Potteiger J, Sullivan DK, Johnson SL, Heelan K, Hise M, Fennessey PV, Sonko B, Sharp T, Jakicic JM, Blair SN, Tran ZV, Mayo M, Gibson C, Washburn RA. Effects of a 16-month randomized controlled exercise trial on body weight and composition in young, overweight men and women: the Midwest Exercise Trial. Arch Intern Med. 2003 Jun 9;163(11):1343-50. doi: 10.1001/archinte.163.11.1343. PMID 12796071
- [Background] Rejeski WJ, Brubaker PH, Goff DC Jr, Bearon LB, McClelland JW, Perri MG, Ambrosius WT. Translating weight loss and physical activity programs into the community to preserve mobility in older, obese adults in poor cardiovascular health. Arch Intern Med. 2011 May 23;171(10):880-6. doi: 10.1001/archinternmed.2010.522. Epub 2011 Jan 24. PMID 21263080
- [Background] Almeida FA, You W, Harden SM, Blackman KC, Davy BM, Glasgow RE, Hill JL, Linnan LA, Wall SS, Yenerall J, Zoellner JM, Estabrooks PA. Effectiveness of a worksite-based weight loss randomized controlled trial: the worksite study. Obesity (Silver Spring). 2015 Apr;23(4):737-45. doi: 10.1002/oby.20899. Epub 2015 Feb 12. PMID 25678325
- [Background] Estabrooks PA, Glasgow RE. Translating effective clinic-based physical activity interventions into practice. Am J Prev Med. 2006 Oct;31(4 Suppl):S45-56. doi: 10.1016/j.amepre.2006.06.019. PMID 16979469
- [Background] Akers JD, Estabrooks PA, Davy BM. Translational research: bridging the gap between long-term weight loss maintenance research and practice. J Am Diet Assoc. 2010 Oct;110(10):1511-22, 1522.e1-3. doi: 10.1016/j.jada.2010.07.005. PMID 20869490
- [Background] Green LW, Glasgow RE, Atkins D, Stange K. Making evidence from research more relevant, useful, and actionable in policy, program planning, and practice slips "twixt cup and lip". Am J Prev Med. 2009 Dec;37(6 Suppl 1):S187-91. doi: 10.1016/j.amepre.2009.08.017. No abstract available. PMID 19896017
- [Background] AuYoung M, Linke SE, Pagoto S, Buman MP, Craft LL, Richardson CR, Hutber A, Marcus BH, Estabrooks P, Sheinfeld Gorin S. Integrating Physical Activity in Primary Care Practice. Am J Med. 2016 Oct;129(10):1022-9. doi: 10.1016/j.amjmed.2016.02.008. Epub 2016 Mar 4. PMID 26953063
- [Background] Chan L, Hart LG, Goodman DC. Geographic access to health care for rural Medicare beneficiaries. J Rural Health. 2006 Spring;22(2):140-6. doi: 10.1111/j.1748-0361.2006.00022.x. PMID 16606425
- [Background] Huang TT-K, Grimm B, Hammond RA. A systems-based typological framework for understanding the sustainability, scalability, and reach of childhood obesity interventions. Child Heal Care. 2011;40(3):253-266. doi:10.1080/02739615.2011.590399
- [Background] Leeman J, Calancie L, Kegler MC, Escoffery CT, Herrmann AK, Thatcher E, Hartman MA, Fernandez ME. Developing Theory to Guide Building Practitioners' Capacity to Implement Evidence-Based Interventions. Health Educ Behav. 2017 Feb;44(1):59-69. doi: 10.1177/1090198115610572. Epub 2016 Jul 10. PMID 26500080
- [Background] Cancer Prevention and Control Research Network. Putting Public Health Evidence in Action. Produced by the Centers for Disease Control and Prevention and the National Cancer Institute. Retreived from http://cpcrn.org/pub/evidence-in-action/, October 2017.
- [Background] Chorpita BF, Daleiden EL, Weisz JR. Identifying and selecting the common elements of evidence based interventions: a distillation and matching model. Ment Health Serv Res. 2005 Mar;7(1):5-20. doi: 10.1007/s11020-005-1962-6. PMID 15832690
- [Background] Leeman J, Calancie L, Hartman MA, Escoffery CT, Herrmann AK, Tague LE, Moore AA, Wilson KM, Schreiner M, Samuel-Hodge C. What strategies are used to build practitioners' capacity to implement community-based interventions and are they effective?: a systematic review. Implement Sci. 2015 May 29;10:80. doi: 10.1186/s13012-015-0272-7. PMID 26018220
- [Background] Wilson KE, Harden SM, Almeida FA, You W, Hill JL, Goessl C, Estabrooks PA. Brief self-efficacy scales for use in weight-loss trials: Preliminary evidence of validity. Psychol Assess. 2016 Oct;28(10):1255-1264. doi: 10.1037/pas0000249. Epub 2015 Nov 30. PMID 26619093
- [Derived] Porter G, Michaud TL, Schwab RJ, Hill JL, Estabrooks PA. Reach Outcomes and Costs of Different Physician Referral Strategies for a Weight Management Program Among Rural Primary Care Patients: Type 3 Hybrid Effectiveness-Implementation Trial. JMIR Form Res. 2021 Oct 20;5(10):e28622. doi: 10.2196/28622. PMID 34668873